CLINICAL TRIAL: NCT05345925
Title: Pressure-Volume (PV) Measurements for Evaluating Cardiac Parameters Using BackBeat Medical's Cardiac Neuromodulation Therapy (CNT) Pacing Signals in Different Physiological Pacing Sites: An Acute Study
Brief Title: PV Loops With CNT in Multiple Pacing Sites
Acronym: CS-07
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: CD Leycom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BBM PV-PHYS CS-07
Record Dates: First submitted 2022-04-08; First posted 2022-04-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Bradycardia; A-V Block
MeSH Terms: conditions — Bradycardia; Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Eligible subjects instrumented for CNT testing
  Interventions: Device: Moderato

INTERVENTIONS:
Device: Moderato — Several algorithms comprising CNT will be delivered by the Moderato Implantable Pulse Generator. Each application will last approximately 3 min with 2 minutes baseline (regular pacing) between them. Hence, each subject will serve as its own control (during pacing) and test (during CNT application). Furthermore, the average control value for the whole group will be compared with the average test values of CNT algorithms at the different ventricular lead locations for efficacy assessments. Stratification of subjects by initial hemodynamic parameters (such as Ejection Fraction, for example) would be possible depending on the total number of subjects in each group.

SUMMARY:
In a multicenter non-randomized acute setting, eligible subjects requiring implant or replacement of an IPG (pacemaker, ICD, CRT-P, CRT-D) will be instrumented to study the effect of CNT from different locations in the RV. CNT effects on BP will be evaluated with a PV conductance catheter in the LV, and with optional BP catheters in the aorta and/or RV. CNT will be delivered by externally by the BackBeat Moderato System IPG.

Abbreviations: CNT, Cardiac Neuromodulation Therapy; IPG, Implanted Pulse Generator; ICD, Implanted Cardiac Defribillator; CRT-P or D, Cardiac Resynchronisation Therapy-Pacemaker or Defibrillator; RV, Right Ventricle; LV, Left Ventricle; BP, Blood Pressure

DETAILED DESCRIPTION:
This will be a multi-center, pilot, open-label, non-randomized acute study. The Moderato System is approved for marketing in Europe (has a CE mark) for standard pacing and the treatment of high blood pressure in patients requiring standard cardiac pacing. The therapy delivered by the Moderato® System is referred to as CNT (Cardiac Neuromodulation Therapy).

This investigation will evaluate the effect of different pacing lead positions on cardiac function and the modulation of the autonomic nervous system using Cardiac Neuromodulation Therapy (CNT) pacing signals. The Study includes both patient who have hypertension and patients that do not have hypertension. Moderato®system is currently not indicated for patients that do not have hypertension.

Subjects indicated for an implant or replacement of a device capable of pacing (pacemaker, ICD, CRT-P, CRT-D) who meet the study inclusion and exclusion criteria may participate in the study and will undergo the following procedure during their device implantation or replacement:

A Right Atrial (RA) lead will be positioned according to standard procedure of the initially planned device implant, or kept in place (in device replacement), or only temporarily introduced and used for the trial procedure. Existing ventricular leads (if any) can be used for the trial procedure, too. The ventricular lead will be temporarily positioned in the different pacing sites according to the following order: RV septal, LBBA, LBB. Pacing and CNT will be performed in each of these sites unless the site is unreachable or pacing is not possible. When trial procedures are finished, the ventricular lead will be positioned according to best practices of the implant or replacement procedure the patient is undergoing. Any lead used temporarily would be removed.

The leads will be connected to a BackBeat Moderato® System IPG, externally to the patient, using a single use, sterile Pacing System Analyzer (PSA) cable provided by the hospital. The Moderato®IPG - which is approved for chronic CNT delivery in hypertensive patients - will function in this trial as a temporary external CNT signal generator for acute application of the therapy; it will not be in direct contact with the subject.

A standard conductance catheter (CD Leycom, The Netherlands) will be introduced through the femoral artery and advanced into the left ventricle to measure cardiac volumes and pressure.

Arterial blood pressure will be measured by introducing a pressure sensor (e.g., Millar catheter) either from another femoral artery sheath or from a radial arterial line.

Right ventricular blood pressure measurements will be taken by introducing a pressure sensor (e.g., Millar catheter) to the right ventricle through an axillary or subclavian sheath.

The Moderato®IPG will be used to generate standard pacing and Cardiac Neuromodulation Therapy (CNT) signals and deliver them to the patient through the cable and leads. A range of CNT signal parameters will be used to assess the effect on sympathetic activity at the different lead positions. Ventricular pressure and volume readings from the conductance catheter, arterial pressure readings and right ventricle pressure readings will be recorded and analyzed to assess the effect of CNT signals on cardiac function, sympathetic activity and blood pressure. The effects of CNT signal over a range of parameter settings will be studied in the different lead positions.

Simultaneous recording of the ventricular and arterial pressures, ventricular volume measurements and ECG signals will be performed in every pacing site during both pacing and CNT using the LEYCOM® Inca (IntraCardiac Analyzer) system, an integrated, stand-alone system for constant monitoring of intra-ventricular pressure and volume (CE marked).

In this study, none of the Moderato® system components will be in contact with the patient. The Moderato® IPG will be used solely as an external CNT signal generator and deliver signals to the patient through the PSA cable and the pacemaker leads.

When CNT signal activation is complete, data recording will be stopped, the conductance catheter will be removed, the cable connecting the IPG to the leads disconnected, and device implantation (or replacement) will proceed normally. Any pacing lead used temporarily would be removed if not required for ongoing patient treatment.

Patients will be considered as having completed the study at the conclusion of the acute procedure unless a safety event is observed during the acute procedure in which case the patients will be followed until the event has been resolved.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject is indicated for an implant or a replacement with a planned upgrade of a device capable of pacing (pacemaker, ICD, CRT-P, CRT-D).
* Subject is willing and able to comply with the study procedures.

Exclusion Criteria:

* Subject is dependent on 100% ventricular pacing.
* Subject has symptoms of heart failure, NYHA Class III or greater
* Subject has an ejection fraction of 25% or less
* Subject's systolic blood pressure is less than 100 mmHg on the day of implant
* Subject has decompensated heart failure
* Subject has significant (>2+) valvular regurgitation or any valvular stenosis.
* Subject has permanent atrial fibrillation
* Subject has atrial fibrillation on the day of the study.
* Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy, or interventricular septal thickness ≥15 mm
* Subject is on dialysis
* Subject has a history of prior neurological events (stroke or TIA) within the past year or a neurological event (stroke) at any prior time that has resulted in residual neurologic deficit.
* Subject has a history of autonomic dysfunction
* Patient cannot receive heparin for any reason (such as a history of Heparin induced thrombocytopenia (HIT))
* Women who are pregnant or breast-feeding
* Subject cannot or is unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-02 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Average changes in Systolic Blood Pressure Change | through study completion (18 months)
  When compared to standard pacing, CNT elicits a reduction in Systolic Blood Pressure (mmHg)

SECONDARY OUTCOMES:
Average Cardiac Volumes (End Diastolic and End Systolic volumes, stroke volumes) | through study completion (18 months)
  When compared to standard pacing, CNT varies cardiac volumes (ml)
Average Ejection Fraction (the percent of blood volume ejected per beat) | through study completion (18 months)
  When compared to standard pacing, CNT varies Ejection Fraction (EF, %)
Average Cardiac Pressures (End Systolic and Diastolic Pressures) | through study completion (18 months)
  When compared to standard pacing, CNT varies cardiac pressures (mmHg)
Average cardiac contractility | through study completion (18 months)
  When compared to standard pacing, CNT varies cardiac contractility (mmHg/sec)
Average Systemic Vascular Resistance | through study completion (18 months)
  When compared to standard pacing, CNT Systemic Resistance (ml/mmHg/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Jastrzębski,, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- University Hospital, Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klotz S, Dickstein ML, Burkhoff D. A computational method of prediction of the end-diastolic pressure-volume relationship by single beat. Nat Protoc. 2007;2(9):2152-8. doi: 10.1038/nprot.2007.270. PMID 17853871
- [Result] Neuzil P, Merkely B, Erglis A, Marinskis G, de Groot JR, Schmidinger H, Rodriguez Venegas M, Voskuil M, Sturmberger T, Petru J, Jongejan N, Aichinger J, Kamzola G, Aidietis A, Geller L, Mraz T, Osztheimer I, Mika Y, Evans S, Burkhoff D, Kuck KH; BackBeat Study Investigators. Pacemaker-Mediated Programmable Hypertension Control Therapy. J Am Heart Assoc. 2017 Dec 23;6(12):e006974. doi: 10.1161/JAHA.117.006974. PMID 29275370
- [Result] Yang B, Wang Y, Zhang F, Ju W, Chen H, Mika Y, Aviv R, Evans SJ, Burkhoff D, Wang J, Chen M. Rationale and evidence for the development of a durable device-based cardiac neuromodulation therapy for hypertension. J Am Soc Hypertens. 2018 May;12(5):381-391. doi: 10.1016/j.jash.2018.03.004. Epub 2018 Mar 21. PMID 29628351
- [Result] Kalarus Z, Merkely B, Neuzil P, Grabowski M, Mitkowski P, Marinskis G, Erglis A, Kazmierczak J, Sturmberger T, Sokal A, Pluta S, Geller L, Osztheimer I, Malek F, Kolodzinska A, Mika Y, Evans SJ, Hastings HM, Burkhoff D, Kuck KH. Pacemaker-Based Cardiac Neuromodulation Therapy in Patients With Hypertension: A Pilot Study. J Am Heart Assoc. 2021 Aug 17;10(16):e020492. doi: 10.1161/JAHA.120.020492. Epub 2021 Aug 13. PMID 34387126